CLINICAL TRIAL: NCT04998812
Title: A Phase IV Multicenter, Open-Label Study Evaluating B Cell Levels In Infants Potentially Exposed To Ocrelizumab During Pregnancy
Brief Title: A Study Evaluating B Cell Levels In Infants Potentially Exposed To Ocrelizumab During Pregnancy
Acronym: MINORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: PPD Development, LP (Industry); Laboratory Corporation of America (Industry); Illingworth Research Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MN42988; 2021-000062-14 (EudraCT Number); 2024-510974-25-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2021-08-06; First posted 2021-08-10 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: ocrelizumab, OCREVUS, placental transfer, pregnancy
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Intervention Model Description: 35 pregnant women with singleton pregnancy were enrolled in the study (70 participants in total, including the infants).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregnant Women with CIS or MS (Experimental): Pregnant women with CIS or MS (in line with the locally approved indications) receiving commercial ocrelizumab up to 6 months before the LMP or during the first trimester of pregnancy (up to gestational week 13), due to accidental exposure, or in whom a decision to treat with ocrelizumab was taken as part of routine clinical practice.
  Interventions: Drug: Ocrelizumab
- Infants (No Intervention): Infants born to women receiving commercial ocrelizumab IV either 0-6 months before the LMP or during the first trimester of pregnancy (up to gestational week 13) due to accidental exposure, or in whom a decision to treat with ocrelizumab was taken as part of routine clinical practice were observed up to month 13 of age.

INTERVENTIONS:
Drug: Ocrelizumab — Post-partum dosing and treatment duration are at the discretion of the physicians, in accordance with local clinical practice and local labelling.
  Arms: Pregnant Women with CIS or MS

SUMMARY:
This study will evaluate the potential placental transfer of ocrelizumab in pregnant women with clinically isolated syndrome (CIS) or multiple sclerosis (MS) [in line with the locally approved indications] whose last dose of ocrelizumab was administered any time from 6 months before the last menstrual period (LMP) through to the first trimester (up to gestational week 13) of pregnancy, and the corresponding pharmacodynamic effects (B cell levels) in the infant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS or CIS (in line with the locally approved indications)
* Currently pregnant with singleton pregnancy at gestational week ≤30 at enrolment
* Documentation that first and second obstetric ultrasound has been conducted before enrolment during the screening period
* Documentation that the last exposure to ocrelizumab occurred up to 6 months before the LMP before the woman became pregnant OR during the first trimester of pregnancy

Exclusion Criteria:

* Last exposure to ocrelizumab >6 months before the woman's LMP or later than the first trimester of pregnancy
* Gestational age at enrolment >30 weeks
* Non-singleton pregnancy
* Received the last dose of ocrelizumab at a different posology other than per the local prescribing information
* Lack of access to ultrasound pre-natal care as part of standard clinical practice
* Prior or current obstetric/gynecological conditions associated with adverse pregnancy outcomes
* Pre-pregnancy body mass index >35 kg/m2
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* Prior or current history of primary or secondary immunodeficiency, or woman in an otherwise severely immunocompromised state
* Significant and uncontrolled disease that may preclude a woman from participating in the study
* Women with known active malignancies or being actively monitored for recurrence of malignancy including solid tumors and hematological malignancies
* Prior or current history of alcohol or drug abuse, or current use of tobacco
* Positive screening tests for hepatitis B
* Treatment with drugs known to have teratogenic effects
* Planned treatment with interferons, glatiramer acetate, or pulsed corticosteroids as a bridging therapy after the last ocrelizumab dose and throughout pregnancy
* Treatment with disease-modifying therapies for MS within their respective half-lives prior to the last ocrelizumab dose or prior to the LMP
* Treatment with natalizumab within 12 weeks prior to the LMP
* Treatment with teriflunomide within the last two years, unless measured plasma concentrations are <0.02 mg/L. If levels are >0.02 mg/L or not known, an accelerated elimination procedure is required
* Treatment with any investigational agent within 6 months or five half-lives of the investigational drug prior to the last ocrelizumab dose or prior to the LMP

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2025-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
- France (2):
  - Hopital Pierre Wertheimer - Hopital Neurologique, Bron
  - Hôpital de la Pitié Salpétrière, Paris
- Germany (3):
  - St. Josef Hospital GmbH, Bochum
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - MultipEL Studies - Institut für klinische Studien, Hamburg
- Hosp. Clinico San Carlos, Madrid, Spain
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 pregnant women (with singleton pregnancy) were enrolled in the study across 10 centers in the United States, Germany, France, Switzerland and Spain. An Informed Consent Form (ICF) for participation of the maternal subject and her unborn was signed and dated by the subject. Where applicable, the written ICF with respect to the infant was also signed and dated by the holder of parental rights as designated by the maternal subject. The study is still ongoing.
Pre-assignment Details: Pregnant women with clinically isolated syndrome (CIS) or multiple sclerosis (MS) who were exposed accidentally or as part of routine clinical practice to commercial ocrelizumab up to 6 months before the last menstrual period (LMP) or during the first trimester of pregnancy were enrolled & potential placental transfer of ocrelizumab in infants was observed.
Groups:
- Women: Pregnant women receiving commercial ocrelizumab intravenously (IV) either 0-6 months before the LMP or during the first trimester of pregnancy (up to gestational week 13) due to accidental exposure, or in whom a decision to treat with ocrelizumab was taken as part of routine clinical practice were enrolled. Ocrelizumab was not administered after enrollment in the study until the infant's birth.
- Infants: Infants born to women receiving commercial ocrelizumab IV either 0-6 months before the LMP or during the first trimester of pregnancy (up to gestational week 13) due to accidental exposure, or in whom a decision to treat with ocrelizumab was taken as part of routine clinical practice were observed until the last visit which was at 1 month (+ 30 days) after the first dose of measles, mumps, and rubella (MMR) vaccine (if first dose is administered at 11 months of age or later) or 1 month (+ 30 days) after second dose of MMR vaccine (if first dose is administered before 11 months of age), or at Month 13 of chronological age (+ 30 days) if MMR vaccine is not planned to be administered.
Period: Pregnancy and Early Post-Partum Period
Arm/Group | Women | Infants
Started | 35 | 35
Subject Gave Birth/Infant Was Born | 35 | 35
Completed | 33 | 34
Not Completed | 2 | 1
Not completed — Participant switches to another treatment of MS | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 0 | 1
Period: Vaccination Period
Arm/Group | Women | Infants
Started | 33 | 34
Completed | 10 | 11
Not Completed | 23 | 23
Not completed — Ongoing in study | 23 | 23

BASELINE CHARACTERISTICS:
Population: Full analysis set women (FASW) included all enrolled pregnant women who were exposed to ocrelizumab either 0-6 months before the LMP or in the first trimester of pregnancy. Full analysis set infants (FASI) included all infants born to women in the FASW who were potentially exposed to ocrelizumab during pregnancy. As consent for race and ethnicity was not obtained, this data has not been reported.
Groups:
- Women: Pregnant women receiving commercial ocrelizumab IV either 0-6 months before the LMP or during the first trimester of pregnancy (up to gestational week 13) due to accidental exposure, or in whom a decision to treat with ocrelizumab was taken as part of routine clinical practice were enrolled. Ocrelizumab was not administered after enrollment in the study until the infant's birth.
- Total: Total of all reporting groups
Arm/Group | Women | Infants | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Customized [Count of Participants; unit: Participants]
  Preterm newborn infants (gestational age <37 weeks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 35 | 35
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 35 | 0 | 35
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 22 | 57
  Male | 0 | 13 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not reported | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Infants With B Cell Levels (Cluster of Differentiation 19 [CD19+] Cells) Below the Lower Limit of Normal (LLN)
Description: The event rate (percentage of infants with B cell levels below LLN) and corresponding Clopper Pearson 95% CI were reported. B-cell reference ranges by week of life (absolute counts) are defined by Borriello et al. 2022.
Time Frame: At Week 6 of infant's life
Population: FASI included all infants born to women in the FASW who were potentially exposed to ocrelizumab during pregnancy. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Infants
Number analyzed (Participants) | 34
percentage of participants | 0 [0 to 10.28]

2. Secondary Outcome: Absolute CD19+ B Cell Count in the Infant Potentially Exposed to Ocrelizumab During Pregnancy
Time Frame: At Week 6 of infant's life
Population: as for outcome 1
Measure: Median (Full Range); unit: cells per microliter (cells/µL)
Arm/Group | Infants
Number analyzed (Participants) | 34
cells per microliter (cells/µL) | 1170.00 [269.0 to 2408.0]

3. Secondary Outcome: Percentage of CD19+ B Cell in the Infant Potentially Exposed to Ocrelizumab During Pregnancy
Time Frame: At Week 6 of infant's life
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of cells
Arm/Group | Infants
Number analyzed (Participants) | 34
percentage of cells | 19.20 [5.2 to 35.3]

4. Secondary Outcome: Serum Concentration of Ocrelizumab in the Umbilical Cord Blood at Birth
Description: Serum ocrelizumab concentrations were measured in the umbilical cord blood at birth (within 1 hour after delivery) to evaluate whether there was placental transfer of ocrelizumab from the mother to the infant. At delivery, blood samples from the umbilical cord were collected. Ocrelizumab serum concentration below the lower limit of quantification (LLOQ =156 ng/ml) was set to zero.
Time Frame: Within 1 hour after delivery (at birth Day 1)
Population: FASI included all infants born to women in the FASW who were potentially exposed to ocrelizumab during pregnancy.
Measure: Median (Full Range); unit: nanograms/milliliter (ng/mL)
Arm/Group | Infants
Number analyzed (Participants) | 35
nanograms/milliliter (ng/mL) | 0.00 [0.0 to 694.0]

5. Secondary Outcome: Serum Concentration of Ocrelizumab in the Infant at Week 6 of Life
Description: Serum ocrelizumab concentrations were measured were measured at 6 weeks of the infants life to evaluate whether there was placental transfer of ocrelizumab from the mother to the infant. Serum samples from the infant were collected.
Time Frame: At Week 6 of infant's life
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Infants
Number analyzed (Participants) | 33
ng/mL | 0.00 [0.0 to 263.0]

6. Secondary Outcome: Serum Concentration of Ocrelizumab in the Mother
Description: Serum concentration of ocrelizumab in the mother during pregnancy (time frame of blood sampling: Week 24-30, Week 35) and at delivery (time frame of blood sampling: within 24 hours after delivery). Ocrelizumab serum concentration below the lower limit of quantification (LLOQ =156 ng/ml) was set to zero.
Time Frame: Baseline (gestational Weeks 24-30), gestational Week 35, and at delivery (within 24 hours after delivery) (at birth Day 1)
Population: FASW included all enrolled pregnant women who were exposed to ocrelizumab either 0-6 months before the LMP or in the first trimester of pregnancy. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Women
Number analyzed (Participants) | 35
ng/mL
  Baseline - Gestational Weeks 24-30 | 0.00 [0.0 to 9090.0]
  Gestational Week 35: number analyzed (Participants) | 34
  Gestational Week 35 | 0.00 [0.0 to 787.0]
  At Delivery | 0.00 [0.0 to 382.0]

7. Secondary Outcome: Percentage of Infants With Adverse Events
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: Up to 17 months
Reporting Status: Not Posted

8. Secondary Outcome: Percentage of Mothers With Adverse Events
Description: as for outcome 7
Time Frame: Up to 17 months
Reporting Status: Not Posted

9. Secondary Outcome: Infant Characteristics at Birth: Body Weight
Description: Day 1 refers to the time an infant's birth.
Time Frame: At birth (Day 1)
Population: FASI included all infants born to women in the FASW who were potentially exposed to ocrelizumab during pregnancy.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Infants
Number analyzed (Participants) | 35
kilogram (kg) | 3.46 (0.43)

10. Secondary Outcome: Infant Characteristics at Birth: Head Circumference
Description: Day 1 refers to the time an infant's birth.
Time Frame: At birth (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeter (cm)
Arm/Group | Infants
Number analyzed (Participants) | 30
centimeter (cm) | 35.08 (1.15)

11. Secondary Outcome: Infant Characteristics at Birth: Body Length
Description: Day 1 refers to the time an infant's birth.
Time Frame: At birth (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Infants
Number analyzed (Participants) | 33
cm | 51.58 (2.15)

12. Secondary Outcome: Percentage of Pregnancies Resulting in Live Births, Therapeutic Abortions, or Stillbirth
Description: Pregnancy outcomes analysed included live births (term and preterm, presence of congenital anomalies) and elective/therapeutic abortions and stillbirths.
Time Frame: During pregnancy (anytime between 37 to 42 weeks of gestation) and at birth (at Day 1)
Population: Safety analysis set women (SAFW) included all enrolled pregnant women who were exposed to ocrelizumab either 0-6 months before the LMP or in the first trimester of pregnancy.
Measure: Number; unit: percentage of pregnancies
Arm/Group | Women
Number analyzed (Participants) | 35
percentage of pregnancies
  Live Births | 100
  Congenital Anomalies | 8.6
  Therapeutic Abortions | 0
  Stillbirth | 0
  Preterm | 0

13. Secondary Outcome: Mean Titers of Antibody Immune Responses to Measles, Mumps, and Rubella (MMR) Vaccination
Description: The immune response to MMR vaccine will be assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine is not planned to be administered. This is to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

14. Secondary Outcome: Percentage of Infants With Positive Humoral Response to MMR Vaccination
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) will be presented for each immunoglobulin G (IgG) antibody titer. Seroprotective titer based on vaccine tests for MMR vaccine are as follows: Anti-Measles Vir IgG(-70)CL: ≥ 120 milli-international units/milliliter (mIU/mL); Anti-MumpsAT Vir iGG(-70)CL: ≥ 17 units per milliliters (U/mL); Anti-Rub Vir IgG(-70)RUOCL: ≥ 10 international units/milliliters (IU/mL).
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

15. Secondary Outcome: Mean Titers of Antibody Immune Responses to Diphtheria-Tetanus-Pertussis (DTP) Vaccine
Description: The immune response to DTP vaccine will be assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine is not planned to be administered. This is to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

16. Secondary Outcome: Percentage of Infants With Positive Humoral Response to DTP Vaccine
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) will be presented for each IgG antibody titer. Seroprotective titer based on vaccine tests for DTP vaccine are as follows: Anti-Diphtheria IgG(-70)CL and Anti-Tetanus Toxoid IgG(-70)RUO: ≥ 0.01 IU/mL; Bordetella pertussis antibodies, IgG: > 1.04 cut-off index (COI).
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

17. Secondary Outcome: Mean Titers of Antibody Immune Responses to Haemophilus Influenzae Type B (Hib) Vaccine
Description: The immune response to Hib vaccine will be assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine is not planned to be administered. This is to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

18. Secondary Outcome: Percentage of Infants With Positive Humoral Response to Hib Vaccine
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) will be presented for each IgG antibody titer. Seroprotective titer based on vaccine tests for Hib vaccine are as follows: Hib, IgG: ≥ 0.15 µg/mL.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

19. Secondary Outcome: Mean Titers of Antibody Immune Responses to Hepatitis B Vaccine (HBV)
Description: The immune response to HBV vaccine will be assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine is not planned to be administered. This is to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

20. Secondary Outcome: Percentage of Infants With Positive Humoral Response to HBV
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) will be presented for each IgG antibody titer. Seroprotective titer based on vaccine tests for HBV vaccine are as follows: Anti-HBs: ≥ 10 mIU/mL.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

21. Secondary Outcome: Mean Titers of Antibody Immune Responses to 13-valent Pneumococcal Conjugate Vaccine (PCV-13)
Description: The immune response to PCV-13 vaccine will be assessed 1 month after the first dose of MMR vaccine (if the first dose is administered at 11 months of age or later) or 1 month after the second dose of MMR vaccine (if the first dose is administered before 11 months of age), or at Month 13 of chronological age if MMR vaccine is not planned to be administered. This is to evaluate whether infants can mount humoral immune responses to clinically relevant vaccines.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

22. Secondary Outcome: Percentage of Infants With Positive Humoral Response to PCV-13
Description: Percentage of infants with positive humoral response (seroprotective titers as defined for the individual vaccine) will be presented for each IgG antibody titer. Seroprotective titer based on vaccine tests for PCV-13 vaccine are as follows: 13 Valent anti-pneumococcal antibody panel: ≥ 0.35 µg/mL.
Time Frame: Up to 1 month after the first or second dose of MMR vaccine (at approximately Month 13)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Mothers: Up to approximately 79 weeks; Infants: Up to approximately 66 weeks
Description: Safety analysis was performed on the safety populations of women (SAFW) and infants (SAFI) separately. The study is still ongoing and data collected up to primary completion date is reported here. Adverse event data will be updated one year after study completion date.
Arm/Group | Women | Infants
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 6/35 | 4/35
Other Adverse Events (participants affected / at risk) | 22/35 | 22/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women (N=35) | Infants (N=35)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neonatal infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 0 (0) | 1 (1)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Uterine inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women (N=35) | Infants (N=35)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 3 (4)
Milk allergy (Immune system disorders) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 5 (5)
COVID-19 (Infections and infestations) | 6 (7) | 4 (4)
Conjunctivitis (Infections and infestations) | 2 (2) | 4 (4)
Ear infection (Infections and infestations) | 0 (0) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (6) | 6 (6)
Sinusitis (Infections and infestations) | 2 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (4) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Perineal injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 0 (0)
Blood immunoglobulin G decreased (Investigations) | 2 (2) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT04998812/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT04998812/SAP_001.pdf